CLINICAL TRIAL: NCT01414309
Title: Prospective Evaluation of Heart Failure Patients With Central Sleep Apnea
Status: Terminated | Type: Observational
Why Stopped: Change in company priorities
Sponsor: Respicardia, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: EP 1137
Record Dates: First submitted 2011-08-09; First posted 2011-08-11 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2015-01

CONDITIONS: Central Sleep Apnea; Heart Failure
Keywords: Heart Failure; Central Sleep Apnea; Sleep Disordered Breathing; Cardiac Dysfunction
MeSH Terms: conditions — Sleep Apnea, Central; Heart Failure; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational patients: Heart Failure patients with moderate to severe central sleep apnea

SUMMARY:
Central sleep apnea (CSA) has been associated with increased mortality and primarily occurs in patients with heart failure (HF). The primary purpose of this study is to document the natural progression of moderate to severe CSA in heart failure patients.

DETAILED DESCRIPTION:
This trial is a prospective, non-randomized observational study in heart failure patients with moderate to severe central sleep apnea (CSA).

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to comply with this protocol and has signed an IRB/MEC approved informed consent (as well as Privacy Protection Authorization in the United States)
* Age is greater than or equal to 18 years
* Known recent history of sleep disordered breathing of predominantly central origin, as evidenced by an overnight PSG with EEG and at least 4 hours of recording that was conducted within 60 days of enrollment and demonstrating the following characteristics:
* AHI greater than or equal to 20
* greater than or equal to 50% of classified events of a central nature
* less than 20% of the total AHI comprised of obstructive apnea events
* Diagnosed chronic heart failure, with medications optimized and stable for at least 30 days prior to the screening PSG, or since the date of the earliest test used for baseline, whichever is longer. Optimal medications include: beta blockade, ACE-I or ARB and diuretics unless contraindicated or not considered medically necessary.

Exclusion Criteria:

* Current or intended use of any mask-based therapy for central sleep apnea
* Baseline oxygen saturation less than or equal to 90% on a stable FiO2
* Severe Chronic Obstructive Pulmonary Disease (COPD) (per GOLD classification system)
* History of cerebrovascular accident (CVA), myocardial infarction (MI), coronary artery bypass grafting (CABG) surgery, or percutaneous coronary intervention (PCI), or any cardiac ablation procedure within the 3 months prior to the study
* Unstable angina
* History of primary pulmonary hypertension
* Currently enrolled in a non-observational (ie, interventional) clinical study that could confound the results of this study
* If subject has an implanted cardiac resynchronization device (CRT), it must have been implanted at least 3 months before enrollment; any other device must have been implanted at least 30 days prior to enrollment
* Life expectancy of less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Apnea-hypopnea index and its components | 6 months
  The primary objective of the study is to determine the natural progression of central sleep apnea, using the apnea-hypopnea index (AHI) and its components evaluated at 6 months.

SECONDARY OUTCOMES:
Clinical status associated with sleep disordered breathing | 6 months
  * Epworth Sleepiness Scale
  * Subject Global Assessment
  * Quality of life as measured by Minnesota Living with Heart Failure Questionnaire
  * HF Clinical Composite
  * Six-minute hall walk
  * NYHA Functional Class
  * Echocardiographic measures of structure and function
  * Subject medications

CONTACTS AND LOCATIONS:
Overall Officials: Robin Germany, M.D., Study Director — Respicardia, Inc.
Locations (4):
- United States (3):
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Central MN Heart at St Cloud, Saint Cloud, Minnesota
  - Sleep Therapy & Research Center, Alamo, San Antonio, Texas
- Charite, Campus Virchow-Klinikum, Berlin, Germany

REFERENCES:
- See also: Sponsor's website — http://www.respicardia.com